CLINICAL TRIAL: NCT03240705
Title: Randomised Controlled Trial of Gratitude Reporting vs no Intervention on Well-being of Medical Students During Clerkship
Brief Title: Increasing Medical Student Well-being Through Gratitude Journaling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16.413
Record Dates: First submitted 2017-05-29; First posted 2017-08-07 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Stress, Psychological
Keywords: Stress; Medical education
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The questionnaires will be coded as to not be able to identify study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gratitude journaling (Experimental): Students perform gratitude journaling 3 times per week on a form. This activity consists of writing elements of their day that brought happiness to them. Can be in keyword form or in sentences.
  Interventions: Behavioral: Gratitude journaling
- No intervention (No Intervention): Students proceed with their surgical clerkship as is standard in our institution.

INTERVENTIONS:
Behavioral: Gratitude journaling — Gratitude journaling 3 times a week during surgical rotation
  Arms: Gratitude journaling

SUMMARY:
Clerkship causes significant stress to medical students. Some interventions to increase well-being have been described but none have been studied prospectively in this context.

The primary objective of this study is to examine the effects of gratitude journaling on medical clerks' perceived well-being.

Students will be randomised to one of two groups: gratitude journaling or no intervention. The participants of the experimental group will be asked to complete an online gratitude journal 3 times per week and will be compared to the participants in the control group.

The students in both groups will answer a standardised questionnaire evaluating well-being before and after their surgical rotation.

Those randomised to the intervention group will perform gratitude journaling three times a week during their surgical rotation. This activity consists of writing something that made them feel happy during their day.

Those randomised in the control group (no intervention) will proceed with their normal rotation, without additional gratitude journaling.

The main outcome will be evaluated by comparing the well-being at the end of the surgical rotation as evaluated by a composite well-being assessment scale between both groups.

DETAILED DESCRIPTION:
Medical education involves 2 years of rotations in different medical and surgical specialties. These cause significant stress to clerks, in particular during the surgery rotation. In other professional fields, mindfulness techniques have shown only small to moderate effect on mental health compared to the control group.

An alternative approach to increasing well-being is gratitude journaling. A study examining this approach in student populations demonstrated enhanced well-being and life satisfaction.

The primary objective of this study is to examine the effects of gratitude journaling on medical clerks' perceived well-being.

Students will be randomised to one of two groups: gratitude journaling or no intervention. The participants of the experimental group will be asked to complete an online gratitude journal 3 times per week and will be compared to the participants in the control group.

The students in both groups will answer a standardised questionnaire evaluating well-being before and after their surgical rotation.

Those randomised to the intervention group will perform gratitude journaling three times a week during their surgical rotation. This activity consists of writing something that made them feel happy during their day.

Those randomised in the control group (no intervention) will proceed with their normal rotation, without additional gratitude journaling.

The main outcome will be evaluated by comparing the well-being at the end of the surgical rotation as evaluated by a composite well-being assessment scale between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Medical students at the University of Montreal about to begin their surgical clerkship rotation.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Well-being | 6 weeks after enrollment
  Medical student well-being at the end of their surgical rotation. Measured by Perceived Stress Scale (Cohen, 1983)
Well-being | 6 weeks after enrollment
  Medical student well-being at the end of their surgical rotation. Measured by Satisfaction with Life Scale (Diener, 1985)

SECONDARY OUTCOMES:
Well-being before and after comparison | 6 weeks after enrollment in study
  Before and after comparison of well-being by comparing initial and post-intervention questionnaires (Perceived Stress Scale (Cohen, 1983))
Compliance with gratitude journaling | 6 weeks after enrollment in study
  Proportion of empty entries in the student's gratitude journal

CONTACTS AND LOCATIONS:
Overall Officials: Erica Patocskai, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Faculté de Médecine de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Dijk I, Lucassen PLBJ, Akkermans RP, van Engelen BGM, van Weel C, Speckens AEM. Effects of Mindfulness-Based Stress Reduction on the Mental Health of Clinical Clerkship Students: A Cluster-Randomized Controlled Trial. Acad Med. 2017 Jul;92(7):1012-1021. doi: 10.1097/ACM.0000000000001546. PMID 28121650
- [Background] Pettitt BJ. Medical student concerns and fears before their third-year surgical clerkship. Am J Surg. 2005 Apr;189(4):492-6. doi: 10.1016/j.amjsurg.2004.09.017. PMID 15820468
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493